CLINICAL TRIAL: NCT02275767
Title: Histological Evaluation of Healing Following Ridge Preservation Using a Combined Cortical/Cancellous Mineralized Freeze-Dried Bone Allograft
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSC2014-454H
Record Dates: First submitted 2014-10-22; First posted 2014-10-27 (Estimated); Results first posted 2016-05-11 (Estimated); Last update posted 2016-05-11 (Estimated); Status verified 2016-04

CONDITIONS: Alveolar Bone Loss
MeSH Terms: conditions — Alveolar Bone Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Combination 50% cortical/50% cancellous FDBA (Experimental): Ridge preservation with Combination 50% cortical/50% cancellous freeze-dried bone allograft (FDBA)
  Interventions: Device: 50% cortical/50% cancellous FDBA
- 100% cortical FDBA (Active Comparator): Ridge preservation with 100% cortical freeze-dried bone allograft (FDBA)
  Interventions: Device: 100% cortical FDBA
- 100% cancellous FDBA (Active Comparator): Ridge preservation with 100% cortical freeze-dried bone allograft (FDBA)
  Interventions: Device: 100% cancellous FDBA

INTERVENTIONS:
Device: 50% cortical/50% cancellous FDBA — Ridge preservation after tooth extraction using 50% cortical/50% cancellous FDBA
  Arms: Combination 50% cortical/50% cancellous FDBA
Device: 100% cortical FDBA — Ridge preservation after tooth extraction using 100% cortical FDBA
  Arms: 100% cortical FDBA
Device: 100% cancellous FDBA — Ridge preservation after tooth extraction using 100% cancellous FDBA
  Arms: 100% cancellous FDBA

SUMMARY:
The study is a 3-arm, parallel-design, randomized, prospective clinical trial.designed to examine histologic wound healing following ridge preservation using cortical bone allograft, cancellous bone allograft, or a combination of both cortical and cancellous bone allograft. This entire protocol involves procedures that are standard care. All materials are FDA-approved materials being used in an FDA-approved manner. The test group subjects will have extraction sockets grafted with a combination of 50% cortical/50% cancellous FDBA. This test group will be compared to two active control groups - one using 100% cortical FDBA and the other using 100% cancellous FDBA. The null hypothesis is that there will be no significant difference in formation of new vital bone between treatment groups (primary outcome).

Each subject will provide a single non-molar tooth site for study treatment. After tooth extraction, the graft material will be placed and covered by a non-resorbable membrane. Following 18-20 weeks of healing, the dental implant will be place, at which time a core of bone will be removed from the site as part of the preparation for the implant. The core biopsy will then be evaluated for the primary histologic outcome of % vital bone formation and secondary histologic outcome of % residual graft material.

DETAILED DESCRIPTION:
The study is designed to examine histologic wound healing following ridge preservation using cortical bone allograft, cancellous bone allograft, or a combination of both cortical and cancellous bone allograft. This entire protocol involves procedures that are standard care. All materials are FDA-approved materials being used in an FDA-approved manner. The study is a 3-arm, parallel-design, randomized, prospective clinical trial. The test group subjects will have extraction sockets grafted with a combination of 50% cortical/50% cancellous FDBA. This test group will be compared to two active control groups - one using 100% cortical FDBA and the other using 100% cancellous FDBA. The null hypothesis is that there will be no significant difference in formation of new vital bone between treatment groups (primary outcome).

Each subject will provide a single non-molar tooth site for study treatment. After tooth extraction, the graft material will be placed and covered by a non-resorbable membrane. Following 18-20 weeks of healing, the dental implant will be place, at which time a core of bone will be removed from the site as part of the preparation for the implant. The core biopsy will then be evaluated for the primary histologic outcome of % vital bone formation and secondary histologic outcome of % residual graft material.

ELIGIBILITY:
Inclusion Criteria: Patients will be included in this study if they qualify the following inclusion criteria:

* Live within 50 miles from the School of Dentistry, University of Texas Health Science Center at San Antonio
* Are able to attend a minimum of 6 visits over a 4-5 month period, as required by the study protocol
* A single rooted tooth that has been identified as requiring extraction
* Desire a dental implant to replace the missing tooth
* Have adequate restorative space for a dental implant-retained restoration
* Have at least 10mm of alveolar bone height, without impinging on the maxillary sinus or inferior alveolar canal.
* Have a dehiscence of the buccal or lingual bony plate of the tooth socket extending no more than 50% of the total depth of the socket.
* Female patients who have undergone a hysterectomy, tubal ligation, or menopause, and non-pregnant women of child-bearing potential.
* Are nonsmokers or former smokers. Current smokers may only be included if they smoke <10 cigarettes per day

Exclusion Criteria:

* Patients who live more than 50 miles from the School of Dentistry, University of Texas Health Science Center at San Antonio
* Patients who do not meet all the inclusion criteria or who will not cooperate with the required follow-up schedule.
* Patients will are mentally incompetent, prisoners, or pregnant.
* Pregnant women or women intending to become pregnant during the study period.
* Smokers who smoke >10 cigarettes per day
* Clinical and/or radiographic determinations which will preclude inclusion in this study are: Active infection other than periodontitis; Inadequate bone dimensions or restorative space for a dental implant; Presence of a disease entity, condition or therapeutic regimen which decreases probability of soft tissue and bony healing, e.g., poorly controlled diabetes, chemotherapeutic and immunosuppressive agents, autoimmune diseases, history of bisphosphonate use or long-term steroid therapy; Positive medical history of endocarditis following oral or dental surgery.
* Sensitivity or allergy to Bacitracin, Gentamicin, Polymyxin B Sulfate, alcohol and/or surfactants

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2014-10; Primary Completion 2016-03 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian L Mealey, DDS, MS, Principal Investigator — UT Health Science Center at San Antonio, School of Dentistry
Locations (1):
- UT Health Science Center at San Antonio, School of Dentistry, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Demetter RS, Calahan BG, Mealey BL. Histologic Evaluation of Wound Healing After Ridge Preservation With Cortical, Cancellous, and Combined Cortico-Cancellous Freeze-Dried Bone Allograft: A Randomized Controlled Clinical Trial. J Periodontol. 2017 Sep;88(9):860-868. doi: 10.1902/jop.2017.170155. Epub 2017 Apr 28. PMID 28452622

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Combination 50% Cortical/50% Cancellous FDBA | 100% Cortical FDBA | 100% Cancellous FDBA
Started | 22 | 22 | 22
Completed | 20 | 18 | 19
Not Completed | 2 | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Combination 50% Cortical/50% Cancellous FDBA | 100% Cortical FDBA | 100% Cancellous FDBA | Total
Number analyzed (Participants) | 22 | 22 | 22 | 66
Age, Continuous [Mean (Full Range); unit: years] | 54.4 [29 to 72] | 52.6 [30 to 69] | 53.7 [27 to 74] | 53.2 [27 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 13 | 10 | 37
  Male | 8 | 9 | 12 | 29

OUTCOME MEASURES:

1. Primary Outcome: % Vital Bone Formation (Histological)
Description: histologic determination of % vital bone formation 18-20 weeks after ridge preservation surgery
Time Frame: 18-20 weeks after ridge preservation
Measure: Mean (Standard Deviation); unit: percentage of total area
Arm/Group | Combination 50% Cortical/50% Cancellous FDBA | 100% Cortical FDBA | 100% Cancellous FDBA
Number analyzed (Participants) | 20 | 18 | 19
percentage of total area | 26.4 (13.2) | 24.5 (8.6) | 28.8 (14.1)

2. Secondary Outcome: % Residual Graft Material (Histological)
Description: histologic determination of % residual graft material 18-20 weeks after ridge preservation surgery
Time Frame: 18-20 weeks after ridge preservation
Measure: Mean (Standard Deviation); unit: percentage of total area
Arm/Group | Combination 50% Cortical/50% Cancellous FDBA | 100% Cortical FDBA | 100% Cancellous FDBA
Number analyzed (Participants) | 20 | 18 | 19
percentage of total area | 23.4 (12.5) | 28.1 (10.7) | 18.8 (8.4)

ADVERSE EVENTS:
Arm/Group | Combination 50% Cortical/50% Cancellous FDBA | 100% Cortical FDBA | 100% Cancellous FDBA
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/22 | 0/22
Other Adverse Events (participants affected / at risk) | 0/22 | 0/22 | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes